CLINICAL TRIAL: NCT00353691
Title: Glimepiride Versus Metformin as Monotherapy in Pediatric Subjects With Type 2 Diabetes Mellitus: A Single Blind Comparison Study
Brief Title: Glimepiride vs Metformin as Monotherapy in Pediatric Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HOE490_4038
Record Dates: First submitted 2006-07-17; First posted 2006-07-19 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride; Metformin

INTERVENTIONS:
Drug: glimepiride
Drug: metformin

SUMMARY:
To compare the change in glycemic control from baseline to endpoint (last available posttreatment assessment) as measured by HbA1c in pediatric subjects with type 2 diabetes receiving either glimepiride or metformin as monotherapy.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Subjects who had type 2 diabetes treated with diet and exercise only for at least 2 weeks prior to randomization, or who were previously or currently treated with an oral agent and had not responded to diet, exercise, and oral therapy for at least 3 months (documented by an HbA1c >7.5%).
2. Subjects who completed glimepiride pharmacokinetic Study HOE 490/4045 at preselected sites within 3 weeks prior to the screening period were also permitted to enroll.
3. Subjects were required to be negative for islet cell antigen (ICA) and glutamic acid decarboxylase (GAD) autoantibodies and to have a C-peptide level at 90 minutes of ≥ 1.5 ng/mL. The HbA1c was required to be >7.1% at screening and <12.0% on the day of randomization.

EXCLUSION CRITERIA:

Subjects meeting any of the following criteria were not to be included in the study:

1. A history of an acute metabolic complication such as diabetic ketoacidosis within 3 months before screening
2. On insulin therapy, or had received insulin for >6 weeks, 3 months prior to randomization
3. On weight-reduction medication
4. Known hypersensitivity to biguanides, sulfonamides, or insulin
5. Pregnant or lactating females
6. Clinically significant renal (serum creatinine level >1.0 mg/dL) or hepatic disease (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] >2.5 times the upper limits of normal [ULN])
7. GI disorders that may interfere with the absorption of the study drugs
8. Chronic use of medications known to affect glucose levels such as intermittent use of systemic corticosteroids or large dose of inhaled steroids
9. Clinically significant laboratory abnormality on screening laboratory tests or any medical condition that in the opinion of the investigator would affect the outcome of the study
10. History of drug or alcohol abuse
11. Treatment with any investigational product in the last 3 months before study entry
12. History of noncompliance with regard to follow-up medical care
13. Any disease or condition that in the opinion of the investigator and/or sponsor may interfere with completion of the study

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100
Dates: Start 2002-10; Study Completion 2004-11

PRIMARY OUTCOMES:
Change in HbA1c from baseline to Week 24 or last evaluable ontreatment value.

SECONDARY OUTCOMES:
Change in HbA1c from baseline to Week 12
Responder rate, defined as proportion of subjects with HbA1c < 7.0% at Week 24 or last evaluable on-therapy observation
Mean change in fasting SMBG from baseline to each visit at weeks 4, 8, 12, 18 and 24 or last evaluable on-treatment value.
Mean change in fasting plasma glucose (FPG) from baseline to each visit at weeks 4, 8, 12, 18 and 24 or last evaluable on-treatment value.
Percent completers, defined as subjects who continued study medication until completion of all requirements of Visit 6 (Week 18)
Mean change in lipid levels (total cholesterol, HDL cholesterol, LDL cholesterol, and triglycerides) from baseline to Wk 24 or last evaluable on-treatment value.
Mean change in body mass index (BMI) from baseline to Wk 12 and Wk 24 or last evaluable on-treatment value

CONTACTS AND LOCATIONS:
Overall Officials: Karen Barch, B.S., Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States

REFERENCES:
- [Derived] Gottschalk M, Danne T, Vlajnic A, Cara JF. Glimepiride versus metformin as monotherapy in pediatric patients with type 2 diabetes: a randomized, single-blind comparative study. Diabetes Care. 2007 Apr;30(4):790-4. doi: 10.2337/dc06-1554. PMID 17392540